CLINICAL TRIAL: NCT00420056
Title: A Pilot Study Of Pd 0332991 In Patients With Previously Treated Mantle Cell Lymphoma
Brief Title: An Investigational Study Drug, Palbociclib (PD-0332991), Is Being Studied In Patients With Mantle Cell Lymphoma. Patients Must Have Received Prior Treatment(s) For Mantle Cell Lymphoma.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5481002
Record Dates: First submitted 2007-01-05; First posted 2007-01-09 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Lymphoma, Mantle-Cell
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PD-0332991 (Experimental)
  Interventions: Drug: PD-0332991

INTERVENTIONS:
Drug: PD-0332991 — 125 mg, oral, Days 1-21 of a 28-day cycle

SUMMARY:
This is a pilot study evaluating tumor activity using Positron Emission Tomography, which is also known as a "PET scan". This study will assess the safety of using PD-0332991 in patients with mantle cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented MCL.
* Must have received at least one prior therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
* Adequate organ function as outlined in the protocol.

Exclusion Criteria:

* Major surgery, radiation therapy, or systemic therapy within 4 weeks of study enrollment.
* Prior radiation therapy to >25% of the bone marrow (whole pelvis is 25%).
* Uncontrolled brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-05; Primary Completion 2010-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Weill Medical College of Cornell University - New York Presbyterian Hospital, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Leonard JP, LaCasce AS, Smith MR, Noy A, Chirieac LR, Rodig SJ, Yu JQ, Vallabhajosula S, Schoder H, English P, Neuberg DS, Martin P, Millenson MM, Ely SA, Courtney R, Shaik N, Wilner KD, Randolph S, Van den Abbeele AD, Chen-Kiang SY, Yap JT, Shapiro GI. Selective CDK4/6 inhibition with tumor responses by PD0332991 in patients with mantle cell lymphoma. Blood. 2012 May 17;119(20):4597-607. doi: 10.1182/blood-2011-10-388298. Epub 2012 Mar 1. PMID 22383795
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481002

RESULTS

PARTICIPANT FLOW:
Groups:
- PD 0332991: PD 0332991 125 milligram (mg) capsule orally once daily in cycles of continuous dosing for 3 weeks followed by 1-week rest, with no dosing (schedule 3/1) until objective disease progression, withdrawal due to unacceptable toxicity or withdrawal of consent by the participant. Dose was reduced up to PD 0332991 75 mg once daily depending on the type and severity of toxicity encountered and as per investigator's discretion.
Period: Overall Study
Arm/Group | PD 0332991
Started | 17
Completed | 0
Not Completed | 17
Not completed — Objective progression or relapse | 17

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants enrolled in the study who received at least 1 dose of study medication.
Arm/Group | PD 0332991
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Correlation Coefficient Between Change From Baseline in Fluoro-L-thymidine Positron Emission Tomography (FLT-PET) Maximum Standard Uptake Value (SUVmax) and in Phosphorylated Retinoblastoma (Phospho-Rb) Percent Positive Cells at Cycle 1 Day 21
Description: Maximum standard uptake value (SUVmax) was defined as the maximum value attained for the ratio of tissue radioactivity concentration at any time and the injected radioactivity concentration divided by the body weight (in kilogram [kg]). Phosphorylation of retinoblastoma (Rb) protein in the tumor cells, expressed as phospho-Rb percent positive cells, was assessed using Immunohistochemical staining technique. Change from baseline in [(18)F]-FLT-PET SUVmax at Cycle 1 Day 21 and change from baseline in Phospho-Rb percent positive cells at Cycle 1 Day 21 were analyzed. The change values of FLT-PET SUVmax and Phospho-Rb percent positive cells were then correlated. Here, 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Time Frame: Baseline, Cycle 1 Day 21
Population: SUVmax was analyzed using imaging analysis set (participants in FAS who completed baseline [(18)F]-fluorodeoxyglucose PET [FDG-PET] and [(18)F]-FLT-PET, and at least 1 on-treatment [Day 21] PET) and phospho-Rb was analyzed using tumor analysis set (participants in FAS who completed tumor biomarker assessments at baseline and Day 21).
Measure: Number; unit: correlation coefficient
Arm/Group | PD 0332991
Number analyzed (Participants) | 10
correlation coefficient | -0.25034
Statistical Analysis 1: Comparison: PD 0332991; Test type: Superiority or Other; p = 0.4854, Regression, Linear

2. Primary Outcome: Correlation Coefficient Between Change From Baseline in Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) Maximum Standard Uptake Value (SUVmax) and in Phosphorylated Retinoblastoma (Phospho-Rb) Percent Positive Cells at Cycle 1 Day 21
Description: Maximum standard uptake value (SUVmax) was defined as the maximum value attained for the ratio of tissue radioactivity concentration at any time and the injected radioactivity concentration divided by the body weight (in kilogram [kg]). Phosphorylation of retinoblastoma (Rb) protein in the tumor cells, expressed as phospho-Rb percent positive cells, was assessed using Immunohistochemical staining technique. Change from baseline in [(18)F]-FDG-PET SUVmax at Cycle 1 Day 21 and change from baseline in Phospho-Rb percent positive cells at Cycle 1 Day 21 were analyzed. The change values of FLT-PET SUVmax and Phospho-Rb percent positive cells were then correlated. Here, 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Time Frame: Baseline, Cycle 1 Day 21
Population: SUVmax was analyzed using imaging analysis set (participants in FAS who completed baseline [(18)F]-FDG-PET and [(18)F]-FLT-PET, and at least 1 on-treatment [Day 21] PET) and phospho-Rb was analyzed using tumor analysis set (participants in FAS who completed tumor biomarker assessments at baseline and Day 21).
Measure: Number; unit: correlation coefficient
Arm/Group | PD 0332991
Number analyzed (Participants) | 10
correlation coefficient | 0.13551
Statistical Analysis 1: Comparison: PD 0332991; Test type: Superiority or Other; p = 0.7090, Regression, Linear

3. Primary Outcome: Change From Baseline in Maximum Standard Uptake Value (SUVmax) at Cycle 1 Day 21
Description: Maximum standard uptake value (SUVmax) was defined as the maximum value attained for the ratio of tissue radioactivity concentration at any time and the injected radioactivity concentration divided by the body weight (in kilogram [kg]). Change from baseline in SUVmax was assessed using [(18)F]-FLT-PET and [(18)F]-FDG-PET techniques.
Time Frame: Baseline, Cycle 1 Day 21
Population: Imaging analysis set included participants in FAS who completed baseline [(18)F]-FDG-PET and [(18)F]-FLT-PET, and at least 1 on-treatment (Day 21) PET.
Measure: Mean (Standard Deviation); unit: standard uptake value (SUV)
Arm/Group | PD 0332991
Number analyzed (Participants) | 17
standard uptake value (SUV)
  Baseline: FLT-PET | 9.964 (4.929)
  Baseline: FDG-PET | 9.049 (4.654)
  Change at Cycle 1 Day 21: FLT-PET | -4.551 (2.968)
  Change at Cycle 1 Day 21: FDG-PET | -2.271 (2.913)

4. Primary Outcome: Correlation Between Positron Emission Tomography (PET) Response and Progression-Free Survival (PFS)
Description: PET response was defined as complete response (CR) = mean SUVmax same as of background; partial response (PR) = mean SUVmax less than (<) 75 percent (%) of baseline; progressive disease (PD) = mean SUVmax greater than (>) 125% of baseline; stable disease (SD) = mean SUVmax greater than or equal to (>=) 75% of baseline and mean SUVmax less than or equal to (<=) 125% of baseline. PFS was defined as the time from first dose of study medication to the first documentation of objective tumor progression, or to death due to any cause, whichever occurred first. Tumor progression was defined as >50% increase in sum of products of diameters, of dominant nodes and documented non-nodal sites or appearance of new sites of disease.
Time Frame: Baseline, Cycle 1 Day 21 for PET response; Screening until tumor progression or death, assessed on Day 1 of every alternate cycle starting from Cycle 1 up to end of treatment (Day 609) or early withdrawal (if not completed during last 6 weeks) for PFS
Population: Analysis for this outcome measure was not run as there were so few responders.
Arm/Group | PD 0332991
Number analyzed (Participants) | 0

5. Primary Outcome: Correlation Between Positron Emission Tomography (PET) Response and Objective Response (OR)
Description: OR: CR= disappearance of all clinical/radiographic evidence of disease, disease related symptoms and biochemical abnormalities, nodal masses regressed to normal size, if spleen and bone marrow were involved, spleen regressed to normal size and not palpable and clear infiltrate on repeat bone marrow aspiration; PR= dominant nodes decreased by >50% in sum of products of diameters (SPD), no increase in size of other nodes/liver/spleen, lesions regressed by >50% in SPD, no new sites of disease; SD= response <PR and no PD, documented >=1 time after start of therapy, no new sites of disease; PD= >50% increase in SPD of dominant nodes and other nodes or appearance of new sites of disease. PET response: CR= mean SUVmax same as background; PR= mean SUVmax <75% of baseline; PD= mean SUVmax >125% of baseline; SD= mean SUVmax >=75% of baseline but <=125% of baseline. Correlation was reported as conjoint number of participants with PET response at Cycle 1 Day 21 and OR at end of study.
Time Frame: Baseline, Cycle 1 Day 21 for PET response; Screening until tumor progression or death, assessed on Day 1 of every alternate cycle starting from Cycle 1 up to end of treatment (Day 609) or early withdrawal (if not completed during last 6 weeks) for OR
Population: PET response was analyzed using Imaging analysis set and OR was analyzed using response analysis set (all participants enrolled in the study who received at least 1 dose of study medication in cycle 1 and for whom a post-treatment response assessment was completed).
Measure: Number; unit: participants
Arm/Group | PD 0332991
Number analyzed (Participants) | 17
participants
  FLT-PET PR, Objective CR | 1
  FLT-PET PR, Objective PR | 2
  FLT-PET PR, Objective SD | 7
  FLT-PET PR, Objective PD | 4
  FLT-PET PR, Indetermined Objective Response | 1
  FLT-PET SD, Objective PD | 2
  FDG-PET PR, Objective PR | 2
  FDG-PET PR, Objective SD | 3
  FDG-PET PR, Objective PD | 2
  FDG-PET SD, Objective CR | 1
  FDG-PET SD, Objective SD | 4
  FDG-PET SD, Objective PD | 4
  FDG-PET SD, Objective Indetermined Response | 1
Statistical Analysis 1: Comparison: PD 0332991; FLT-PET response versus Objective response; Test type: Superiority or Other; Kappa = 0.0638, 95% CI 2-sided [-0.0449 to 0.1726]
Statistical Analysis 2: Comparison: PD 0332991; FDG-PET response versus Objective response; Test type: Superiority or Other; Kappa = 0.1864, 95% CI 2-sided [-0.2316 to 0.6045]

6. Primary Outcome: Phosphorylated Retinoblastoma (Phospho-Rb) Percent Positive Cells at Baseline
Description: Phosphorylation of retinoblastoma (Rb) protein in the tumor cells, expressed as phospho-Rb percent positive cells, was assessed using Immunohistochemical staining technique.
Time Frame: Baseline
Population: Tumor analysis set include all participants in FAS who completed tumor biomarker assessments at baseline and Day 21. Here, 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: percentage of tumor cells
Arm/Group | PD 0332991
Number analyzed (Participants) | 10
percentage of tumor cells | 47.9 (25.72)

7. Primary Outcome: Phosphorylated Retinoblastoma (Phospho-Rb) Percent Positive Cells at Cycle 1 Day 21
Description: as for outcome 6
Time Frame: Cycle 1 Day 21
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of tumor cells
Arm/Group | PD 0332991
Number analyzed (Participants) | 10
percentage of tumor cells | 7.2 (14.4)

8. Primary Outcome: Ki-67 Composite Score at Baseline
Description: Percentage of Ki-67 positive cells was determined by Immunohistochemical staining technique. Composite score = (sum of each intensity category multiplied by percent of cells in that category). Intensity categories of staining (0 = no staining; 1 = weak staining; 2 = moderate staining; 3 = strong staining). Composite score ranges from 0 (no staining) to 300 (100% of cells with 3 staining intensity).
Time Frame: Baseline
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PD 0332991
Number analyzed (Participants) | 6
units on a scale | 191.2 (64.56)

9. Primary Outcome: Ki-67 Composite Score at Cycle 1 Day 21
Description: as for outcome 8
Time Frame: Cycle 1 Day 21
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PD 0332991
Number analyzed (Participants) | 6
units on a scale | 78.5 (110.02)

10. Primary Outcome: Cyclin D1 Composite Score at Baseline
Description: Percentage of Cyclin D1 positive cells was determined by Immunohistochemical staining technique. Composite score = (sum of each intensity category multiplied by percent of cells in that category). Intensity categories of staining (0 = no staining; 1 = weak staining; 2 = moderate staining; 3 = strong staining). Composite score ranges from 0 (no staining) to 300 (100% of cells with 3 staining intensity).
Time Frame: Baseline
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PD 0332991
Number analyzed (Participants) | 6
units on a scale | 165.0 (78.17)

11. Primary Outcome: Cyclin D1 Composite Score at Cycle 1 Day 21
Description: as for outcome 10
Time Frame: Cycle 1 Day 21
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PD 0332991
Number analyzed (Participants) | 6
units on a scale | 124.2 (47.58)

12. Primary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Criteria for laboratory test abnormality: Hematology (Hemoglobin [<0.8*lower limit of normal {LLN}], Platelets [<0.5*LLN/ >1.75*upper limit of normal {ULN}], White blood cells [<0.6*LLN/ >1.5*ULN], Lymphocytes, Neutrophils [<0.8*LLN/ >1.2*ULN], Basophils, Eosinophils, Monocytes [>1.2*ULN]); Liver Function (Total bilirubin [>1.5*ULN], Aspartate aminotransferase, Alanine aminotransferase, Lactate dehydrogenase, Alkaline phosphatase [>0.3*ULN], Total protein, Albumin [<0.8*LLN/ >1.2*ULN]); Renal Function (Blood urea nitrogen, Creatinine [>1.3*ULN], Uric acid [>1.2*ULN]); Electrolytes (sodium [<0.95*LLN/ >1.05*ULN], potassium, chloride, calcium, magnesium [<0.9*LLN/ >1.1*ULN], phosphate [<0.8*LLN/ >1.2*ULN]); Other (Glucose [<0.6*LLN/ >1.5*ULN]).
Time Frame: Baseline up to 28 days after last dose of study medication
Population: Safety analysis set included all participants enrolled in the study who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PD 0332991
Number analyzed (Participants) | 17
participants | 16

13. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events by Severity
Description: AE = any untoward medical occurrence in participant who received study medication without regard to possibility of causal relationship. Severity was assessed as: Grade 1 (Mild); Grade 2 (Moderate); Grade 3 (Severe) = unacceptable or intolerable events, significantly interrupting usual daily activity, and requiring systemic medication therapy/other treatment; Grade 4 (Life-threatening) = events causing participant to be in imminent danger of death; Grade 5 (Death) = death related to an AE. Treatment-emergent events = between first dose of study medication and up to 28 days after last dose, that were absent before treatment or that worsened relative to pre-treatment state. A participant may be represented in more than 1 category.
Time Frame: Day 1 up to 28 days after last dose of study medication
Population: Safety analysis set included all participants enrolled in the study who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PD 0332991
Number analyzed (Participants) | 17
participants
  Grade 1 | 4
  Grade 2 | 2
  Grade 3 | 7
  Grade 4 | 3
  Grade 5 | 1

14. Primary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The events which were considered treatment-related by sponsor and/or investigator were reported.
Time Frame: Day 1 up to 28 days after last dose of study medication
Population: Safety analysis set included all participants enrolled in the study who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PD 0332991
Number analyzed (Participants) | 17
participants
  AEs | 16
  SAEs | 2

15. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from first dose of study medication to the first documentation of objective tumor progression, or to death due to any cause, whichever occurred first. Tumor progression was defined as >50% increase in sum of products of diameters, of dominant nodes and documented non-nodal sites or appearance of new sites of disease. PFS= (first event date minus the first dose date plus 1) divided by 30.44.
Time Frame: Screening until tumor progression or death, assessed on Day 1 of every alternate cycle starting from Cycle 1 up to end of treatment (Day 609) or early withdrawal (if not completed during last 6 weeks)
Population: Response analysis set included all participants enrolled in the study who received at least 1 dose of study medication in cycle 1 and for whom a post-treatment response assessment was completed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PD 0332991
Number analyzed (Participants) | 16
months | 5.5 [2.0 to 18.6]

16. Secondary Outcome: Percentage of Participants With Objective Response
Description: OR is defined as the percentage of participants with confirmed complete response (CR) or confirmed partial response (PR). Confirmed responses are those that persist on repeat imaging study 4 weeks after initial documentation of response. Complete response (CR)= disappearance of all detectable clinical/radiographic evidence of disease, disease related symptoms present before therapy and biochemical abnormalities attributable to disease, nodal masses regressed to normal size, if spleen and bone marrow were involved, spleen regressed to normal size and not palpable and clear infiltrate on repeated bone marrow aspiration; Partial response (PR)= dominant nodes decreased by >50% in sum of products of diameters (SPD), no increase in size of other nodes/liver/spleen, lesions in organs (spleen/liver) regressed by >50% in SPD, no new sites of disease.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PD 0332991
Number analyzed (Participants) | 16
percentage of participants | 18.8 [4.0 to 45.6]

17. Secondary Outcome: Duration of Response (DR)
Description: Time in months from first documentation of objective tumor response (CR or PR) that was subsequently confirmed, to objective tumor progression (PD) or death due to any cause. DR= (date of first documentation of PD or death, minus the date of first CR or PR plus 1) divided by 30.44. CR= disappearance of all detectable clinical/radiographic evidence of disease, disease related symptoms present before start of therapy and biochemical abnormalities attributable to disease, nodal masses regressed to normal size, if spleen and bone marrow were involved, spleen regressed to normal size and not palpable and clear infiltrate on repeated bone marrow aspiration. PR= dominant nodes decreased by >50% in sum of products of diameters (SPD), no increase in size of other nodes/liver/spleen, lesions in organs (spleen/liver) regressed by >50% in SPD, no new sites of disease. PD= >50% increase in SPD of dominant nodes and other nodes or appearance of new sites of disease.
Time Frame: as for outcome 15
Population: For duration of response, the number of participants experiencing objective response was less than 50%, and therefore, it was not feasible to calculate duration of response using Kaplan-Meier method. Hence, no participant was analyzed for this outcome measure.
Arm/Group | PD 0332991
Number analyzed (Participants) | 0

18. Secondary Outcome: Time to Tumor Progression (TTP)
Description: Time in months from date of first dose of study medication to first documentation of objective tumor progression (PD). TTP= (last known progression-free date minus date of first dose of study medication plus 1) divided by 30.44. PD was defined as greater than 50% increase in sum of products of diameters, of dominant nodes and documented non-nodal sites or appearance of new sites of disease.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PD 0332991
Number analyzed (Participants) | 16
months | 5.5 [2.0 to 18.6]

19. Secondary Outcome: Correlation Coefficient Between Plasma PD 0332991 Concentration and Change From Baseline in Biomarkers and SUVmax at Cycle 1 Day 21
Description: Plasma PD 0332991 concentration at Cycle 1 Day 21 was analyzed. Change from baseline in biomarkers (Ki-67 composite score, Cyclin D1 composite score, phospho-Rb positive cells) and SUVmax (FLT-PET SUVmax, FDG-PET SUVmax) at Cycle 1 Day 21 were analyzed. Correlation between PD 0332991 concentration and change in biomarkers (concentration versus Ki-67, concentration versus Cyclin, and concentration versus phospho-Rb) and SUVmax (concentration versus FLT-PET SUVmax, concentration versus FDG-PET SUVmax) was then assessed. Composite score = (sum of each intensity category multiplied by percent of cells in that category). Intensity categories of staining (0 = no staining; 1 = weak staining; 2 = moderate staining; 3 = strong staining). Here, 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Time Frame: Baseline, Cycle 1 Day 21
Population: PD 0332991 concentration was analyzed using pharmacokinetic analysis set (participants in FAS who had also completed pharmacokinetic blood sampling for at least 1 day); SUVmax and biomarkers were analyzed using imaging analysis set and tumor analysis set respectively. n= participants evaluable for this measure for specified comparisons.
Measure: Number; unit: correlation coefficient
Arm/Group | PD 0332991
Number analyzed (Participants) | 16
correlation coefficient
  Concentration versus Ki-67 (n=6) | 0.27677
  Concentration versus Cyclin D1 (n= 6) | -0.69081
  Concentration versus phospho-Rb (n= 10) | -0.55533
  Concentration versus FLT-PET SUVmax (n= 16) | 0.28767
  Concentration versus FDG-PET SUVmax (n= 16) | -0.18526
Statistical Analysis 1: Comparison: PD 0332991; Concentration versus Ki-67; Test type: Superiority or Other; p = 0.5954, Regression, Linear
Statistical Analysis 2: Comparison: PD 0332991; Concentration versus Cyclin D1; Test type: Superiority or Other; p = 0.1286, Regression, Linear
Statistical Analysis 3: Comparison: PD 0332991; Concentration versus phospho-Rb; Test type: Superiority or Other; p = 0.0956, Regression, Linear
Statistical Analysis 4: Comparison: PD 0332991; Concentration versus FLT-PET SUVmax; Test type: Superiority or Other; p = 0.2800, Regression, Linear
Statistical Analysis 5: Comparison: PD 0332991; Concentration versus FDG-PET SUVmax; Test type: Superiority or Other; p = 0.4921, Regression, Linear

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PD 0332991
Serious Adverse Events (participants affected / at risk) | 3/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PD 0332991 (N=17)
Cardiac arrest (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PD 0332991 (N=17)
Anaemia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 3
Macrocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Palpitations (Cardiac disorders) | 2
Ear pain (Ear and labyrinth disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Vision blurred (Eye disorders) | 2
Visual impairment (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Haematochezia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Axillary pain (General disorders) | 1
Chest pain (General disorders) | 2
Chills (General disorders) | 1
Fatigue (General disorders) | 6
Influenza like illness (General disorders) | 1
Infusion site extravasation (General disorders) | 1
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 2
Thirst (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Balanitis candida (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Proctitis monilial (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Balance disorder (Nervous system disorders) | 1
Brachial plexopathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Hypogeusia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Scrotal pain (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 6
Hot flush (Vascular disorders) | 1
Hypotension (Vascular disorders) | 3
Tympanic membrane perforation (Ear and labyrinth disorders) | 1
Oedema (General disorders) | 1
Eye infection (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Tendon injury (Injury, poisoning and procedural complications) | 1
Blood phosphorus decreased (Investigations) | 1
Hypoaesthesia (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
Results are reported for change from baseline in maximum standard uptake value (SUVmax) instead of percent change from baseline in SUVmax.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.